CLINICAL TRIAL: NCT06789549
Title: Comparing the Efficacy of Epinephrine Nasal Drops and Oxymetazoline Nasal Drops in Reducing Epistaxis During Nasal Intubation: A Randomized Controlled Trial
Brief Title: Epinephrine Nasal Drops for Epistaxis During Nasal Intubation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AN-202501.01
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Oral Surgery
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- epinephrine nasal drops (Experimental): twenty patients was be administered randomly 1 mL of 0.1% epinephrine nasal drops.
  Interventions: Drug: epinephrine nasal drops
- oxymetazoline nasal drops (Active Comparator): twenty patients was be administered randomly receives 1 mL of 0.05% oxymetazoline nasal drops
  Interventions: Drug: oxymetazoline nasal drops

INTERVENTIONS:
Drug: epinephrine nasal drops — Patients in experimental arms received 1 mL of 0.1% epinephrine nasal drops before nasotracheal intubation
  Other Names: Epinephrine 1mg/ml - Pt. Pharos Tbk
  Arms: epinephrine nasal drops
Drug: oxymetazoline nasal drops — Patients in experimental arms received 1 mL of 0.1% oxymetazoline nasal drops before nasotracheal intubation
  Other Names: Oxymetazoline - Iliadin nasal drop 0,05%
  Arms: oxymetazoline nasal drops

SUMMARY:
Epistaxis is the most common complication of nasotracheal intubation. Incidence of epistaxis during nasotracheal intubation ranges from 22% to 80%. Epistaxis during nasotracheal intubation can lead to several complications such as nasal discomfort, airway obstruction, and blood aspiration. The most commonly used and available topical vasoconstrictor in drop form is oxymetazoline. However, oxymetazoline may not always be available in some hospitals, so epinephrine can be used as an alternative nasal decongestant to reduce the incidence of epistaxis during nasotracheal intubation.

DETAILED DESCRIPTION:
Epistaxis associated with nasotracheal intubation can be from blood-tinged mucus to massive bleeding. Epistaxis during nasotracheal intubation can cause excessive force during the procedure, use of an endotracheal tube (ETT) larger than the nasal cavity, repeated intubation attempts, and abnormalities in the anatomy of the nose or nasopharynx. Epistaxis during nasotracheal intubation can lead to several complications such as nasal discomfort, airway obstruction, and blood aspiration.

Topical vasoconstrictors such as oxymetazoline are used to reduce the incidence and severity of epistaxis caused by nasotracheal intubation. Oxymetazoline nasal drops before nasotracheal intubation significantly increases the intranasal diameter and causes vasoconstriction of blood vessels, thereby reducing bleeding and damage to the nasal mucosa.

Epinephrine can be used as an alternative nasal decongestant to reduce the incidence of epistaxis during nasotracheal intubation. Administering 1 mL of 0.1% topical epinephrine reduces 25% nasal mucosal volume and decreases 37% blood flow, thereby providing nasal cavity expansion with lower hemodynamic and systemic effects.

Currently, there exists a lack of empirical research regarding the utilization of epinephrine drops for the prophylaxis of epistaxis in the context of nasotracheal intubation. Given this gap in the literature, the objective of this investigation is to conduct a comparative analysis between the application of 0.1% epinephrine nasal drops and 0.05% oxymetazoline nasal drops for the prevention of epistaxis during nasotracheal intubation procedures for oral surgery.

ELIGIBILITY:
Inclusion Criteria: patients

* underwent oral surgery with nasotracheal intubation
* aged 18-50 years
* ASA (American Society of Anesthesiologists) physical status of 1-2.

Exclusion Criteria:

* allergy to the medications used
* nasal congestion, nasal polyps, allergic rhinitis
* hypertension and use of antihypertensive medications,
* abnormal coagulation factors, receiving antithrombotic and anticoagulant therapy,
* difficult intubation with a LEMON score ≥4,
* a history of nasal surgery or nasal trauma,
* pregnancy,
* heart abnormalities,
* ischemic heart disease or arrhythmias,
* symptoms of acute respiratory infection perioperatively,
* liver and kidney function abnormalities, and
* a history of spontaneous epistaxis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Epistaxis | 2 hour
  The level of epistaxis was assessed during laryngoscopy intubation, 10 minutes after intubation using laryngoscopy, and immediately after extubation.
  The degree of epistaxis was graded on 4 levels:
  None: no bleeding on the posterior pharyngeal wall at the time of intubation and 10 minutes after intubation, and no bleeding from the nasal cavity after extubation.
  Mild: bleeding on the posterior pharyngeal at intubation, no bleeding in the posterior wall of the pharynx 10 minutes after intubation, and no bleeding from the nasal cavity at extubation (bleeding occurs at only one of these times).
  Moderate: bleeding on the posterior pharyngeal at the time intubation and 10 minutes after intubation, but no bleeding from the nasal cavity at extubation (bleeding occurs at two of these times).
  Severe: bleeding on the posterior pharyngeal at the time intubation, 10 minutes after intubation, and bleeding from the nasal cavity at extubation (bleeding occurs at all three times).

SECONDARY OUTCOMES:
Hemodynamic variables | 2 hour
  This outcome reported : Systolic blood pressure (mmHg), diastolic blood pressure (mmHg), MAP (mmHg)
heart rate (bpm) | 2 hour
  Hemodynamic variable

CONTACTS AND LOCATIONS:
Overall Officials: Iwan Fuadi, M.D., PhD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Only resume of demographic and clinical characteristics, included age, height, weight, ASA physical status, gender, ETT size, duration of anesthesia, and duration of surgery, will be shared